CLINICAL TRIAL: NCT06997679
Title: Effects of Continuous Passive Movements Versus Intermittent Compression in Patients With Post ACL Reconstruction Surgery
Brief Title: Effects of Continuous Passive Movements vs Intermittent Compression in Patients With Post ACL Reconstruction Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/825
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving CPM (Experimental)
  Interventions: Diagnostic Test: Patients receiving CPM
- Patients receiving intermittent compression (Active Comparator)
  Interventions: Combination Product: Patients receiving intermittent compression

INTERVENTIONS:
Diagnostic Test: Patients receiving CPM — Group A was treated with Continuous Passive Motion for 30-45 minutes for 2 sessions per day for 8 weeks. CPM can be initiated in the immediate post-operative period, typically within 24-48 hours after surgery. Range of motion will be 0-90 degrees of flexion, with a gradual increase in range over time. Speed is 1-2 cycles per minute. Therapist will Monitor patients for pain and discomfort during CPM, and adjust the protocol as needed. Therapist will Monitor patients range of motion and adjust the CPM protocol to ensure optimal progress. Therapist will monitor patients' knee functions and adjusts the CMP protocol to ensure optimal progress
  Arms: Patients receiving CPM
Combination Product: Patients receiving intermittent compression — Group B was treated with Intermittent Compression Therapy for 30-45 minutes for 2 sessions (morning and evening) per day for 8 weeks. Therapist stand beside the patient .IC therapy initiated in the immediate post-operative period, typically within 24-48 hours after surgery .Pressure of device between 30-40 mmHg and Cycle time is 10-30 seconds inflation, 10-30 seconds deflation. Therapist will Monitor patients for pain and discomfort during IC therapy, and adjust the protocol as needed. Therapist will Monitor patients' swelling and edema, and adjust the IC therapy protocol to ensure optimal progress. Therapist will Monitor patients' knees functions and adjust the IC therapy protocol to ensure optimal progress.
  Arms: Patients receiving intermittent compression

SUMMARY:
ACL Reconstruction Surgery remains a prevalent and debilitating condition, despite invasive and non-invasive approaches aimed at reducing pain and improving function. This study investigates the additional benefits of Continuous Passive Motion (device based exercise) and Intermittent Compression Therapy (device based program) in individuals with Post ACL Reconstruction Surgery.

DETAILED DESCRIPTION:
The researcher employs a randomized controlled trial methodology. Participants are enrolled into two groups: one receiving Continuous Passive Motion (CPM), and the other receiving Intermittent Compression Therapy(IC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by Orthopedic Surgeon and patients who have undergone ACL reconstruction surgery
* Patients who have undergone arthroscopic ACL reconstruction surgery
* Both male and female
* Patients who are within 4th week post-operatively
* Aged between 20-50

Exclusion Criteria:

* Concomitant injuries such as meniscal tears or ligament sprains
* Patients who have undergone previous knee surgery, including ACL reconstruction
* Neurological Condition
* Cardiovascular disease
* Patients with allergies or sensitivities to the materials used in the CPM or IC devices

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale VAS | 12 Months
  The 10-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine" or "worst pain imaginable".
Knee injury and osteoarthritis outcome score KOOS | 12 Months
  The questionnaire has been designed to evaluate Assess the symptoms, function, and quality of life of patients with knee injuries (ACL) or osteoarthritis. There are 5 sections with 42 questions. Each section total score is 100. Each question score between 0-4.Score of 8-10 points is considered clinically significant. Symptoms includes 7 questions which between 0-100. Severe symptoms (0-30), Moderate symptoms (31-60), Mild symptoms (61-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Shalamar Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No